CLINICAL TRIAL: NCT06909162
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Food on the Single-Dose Pharmacokinetics and a Drug-Drug Interaction Evaluation of Itraconazole and Rifampin on INCB123667 When Administered Orally to Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Food on the Single-Dose Pharmacokinetics and a Drug-Drug Interaction Evaluation of Itraconazole and Rifampin on INCB123667 When Administered Orally to Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INCB123667-102
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: INCB123667
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Treatment A - INCB123667 Fasted (Experimental): INCB123667 will be administered at the protocol defined dose.
  Interventions: Drug: INCB123667
- Cohort 1: Treatment B - INCB123667 Fed (Experimental): INCB123667 will be administered at the protocol defined dose.
  Interventions: Drug: INCB123667
- Cohort 2: INCB123667 and itraconazole (Experimental): INCB123667 and itraconazole will be administered at protocol defined doses.
  Interventions: Drug: INCB123667; Drug: itraconazole
- Cohort 3: INCB123667 and rifampin (Experimental): INCB123667 and rifampin will be administered at protocol defined doses.
  Interventions: Drug: INCB123667; Drug: rifampin

INTERVENTIONS:
Drug: INCB123667 — single dose administered orally
Drug: itraconazole — Oral: Tablet
  Arms: Cohort 2: INCB123667 and itraconazole
Drug: rifampin — Oral; Tablet
  Arms: Cohort 3: INCB123667 and rifampin

SUMMARY:
This study will be conducted to evaluate the effect of food on the single-dose pharmacokinetics and a drug-drug interaction evaluation of itraconazole and rifampin on INCB123667 when administered orally to healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Age 19 (in compliance with Nebraska state law) to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening. Note: Only up to 25% of the participants may be enrolled with a BMI > 30 to ≤ 32.0 kg/m2.
* No clinically significant findings on screening evaluations (clinical, laboratory results [with the exception of lipids], and ECGs).
* Ability to swallow and retain oral tablets.
* Willingness to avoid pregnancy or fathering children based on the criteria below:

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children from screening through 90 days (a spermatogenesis cycle) after the last dose of study drug and must refrain from donating sperm during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in on Day -1 and must agree to take appropriate precautions to avoid pregnancy from screening through 30 days (1 menstrual cycle) after the last dose of study drug and must refrain from donating oocytes during this period. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants not considered to be of childbearing potential as defined in the protocol are eligible.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of an autoimmune disease diagnosis (i.e., myasthenia gravis).
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg at screening, confirmed by repeat testing).
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant. Participants with a QTcF interval > 470 milliseconds (females) and > 450 milliseconds (males), QRS interval > 120 milliseconds, or PR interval > 220 milliseconds will be excluded. In the event a value is exclusionary, a single ECG will be repeated twice, and an average taken of the 3 readings will be used to determine if a participant should be excluded.
* Presence or history of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn's disease or chronic pancreatitis).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy; excluding appendectomy and hernia repair) that could affect the absorption of study drug.
* Confirmed resting pulse rate (up to 2 consecutive measurements) < 40 bpm or > 100 bpm at screening.
* Hemoglobin (11.1-15.9 g/dL), WBC (3.4-10.8 / μL), platelet count, or absolute neutrophil count (1.4-7.0 / μL) less than the laboratory LLN at screening or at check-in, confirmed by repeat testing. White blood cell, hemoglobin, neutrophil, and platelet abnormalities must also be clinically significant in the opinion of the investigator to be exclusionary.
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening or at each check-in, confirmed by repeat testing (except participants with Gilbert's disease, for whom total bilirubin must be ≤ 2.0 × ULN).
* Estimated glomerular filtration rate < 90 mL/min / 1.73 m2 based on the site's standard formula at screening (eGFR [mL/min] = eGFR [mL/min / 1.73m2] × [body surface area / 1.73]).

NOTE: Assessment of eGFR may be repeated once if outside of the reference range.

* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Blood transfusion within 4 months of check-in (Day -1).
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes latent treated tuberculosis).
* Known tuberculosis infection that is active or participant-reported history of tuberculosis or treatment thereof.
* Positive test result for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* Receipt of live (including attenuated) vaccines or anticipation of need for such a vaccine during the study.

Note: No vaccines of any type may be administered within 3 months prior to the first dose of study treatment.

* Medical or self-reported history of alcoholism within 3 years of screening.
* History of significant alcohol use within 3 months of screening, defined as regular alcohol consumption > 21 units per week for males and > 14 units for females (1 unit = 0.5 pint beer or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
* Positive urine or breath test result for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 15 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of CYP3A4, P-gp, or breast cancer resistance protein (refer to the Certara Drug Interaction Database Program for prohibited drugs [Certara Drug Interaction Solutions]).
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 72 hours before the first dose of study drug.
* Current use of prohibited medication as described in the protocol.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to INCB123667 or any excipients of INCB123667 or any CDK2 inhibitors.
* Inability to undergo venipuncture or tolerate venous access. Participant has inadequate veins for repeat venipuncture or venous access as determined by the investigator.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* History of tobacco or nicotine-containing product use within 1 month of screening.
* Use of prescription drugs (including hormonal contraceptives) within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days of study drug administration. However, occasional and standard-dose acetaminophen, ibuprofen, and standard-dose vitamins are permitted. Mega dose vitamins or supplements are not permissible.
* Women who are pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Excessive exercise (eg, Ironman, bi/triathlon) within the last 3 months.
* Vitamin B12, folate, TSH, or parathyroid hormone levels less than the laboratory LLN at screening that are clinically significant in the opinion of the investigator.
* Participants with laboratory values outside the normal range at screening as (see protocol for required laboratory analytes). Participants with out-of-range values will be assessed by the investigator or designee for eligibility.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter (PK): Cmax of INCB123667 | Up to Day 16
  Defined as the maximum observed plasma or serum concentration.
Pharmacokinetics Parameter: Tmax of INCB123667 | Up to Day 16
  Defined as the time to maximum concentration.
Pharmacokinetics Parameter: AUCt of INCB123667 | Up to Day 16
  Defined as the area under the steady-state plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Pharmacokinetics Parameter: AUC∞ of INCB123667 | Up to Day 16
  Defined as the area under the single-dose plasma or serum concentration-time curve extrapolated to time of infinity.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 45
  Defined as AEs reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Pharmacokinetics Parameter: tmax of INCB123667 | Up to Day 16
  Defined as the time to maximum concentration.
Pharmacokinetics Parameter: t½ of INCB123667 | Up to Day 16
  Defined as the apparent terminal-phase disposition half-life.
Pharmacokinetics Parameter: CL/F of INCB123667 | Up to Day 16
  Defined as the apparent oral dose clearance.
Pharmacokinetics Parameter: Vz/F of INCB123667 | Up to Day 16
  Defined as the apparent oral dose volume of distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Effect of Food on the Single-Dose Pharmacokinetics of INCB123667 When Administered Orally to Healthy Adult Participants — https://www.incyteclinicaltrials.com/trials/INCB123667-102